CLINICAL TRIAL: NCT03878615
Title: Inflammation and Organ Impact During Hepatic Surgery
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ellinor Wisén, MD, consultant, Sahlgrenska University Hospital
Other Study IDs: Dnr740-18
Record Dates: First submitted 2018-11-06; First posted 2019-03-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Surgery
Keywords: liver surgery; hepatic resection; inflammation; organ dysfunction; blood loss; IFABP
MeSH Terms: conditions — Inflammation; Hemorrhage | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and urinary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Hepatic Surgery: Patientes undergoing elective hepatic resection, managed according to departement routine.
  Interventions: Procedure: elective surgery, according to deprtement routine

INTERVENTIONS:
Procedure: elective surgery, according to deprtement routine — none, descriptive study

SUMMARY:
Monitoring of inflammatory substances (such as interleukins, CRP, albumine), and markers of organ dysfunction (such as creatinine, proenkephaline, amylase, troponine, IFABP and lactate) during elective liver resection. The study also includes monitoring of hemodynamic parameters, blood loss and postoperative complications. Results are to be used för power calculation for future trials.

DETAILED DESCRIPTION:
During hepatic surgery, blood and urine samples will be obtained at 3 times during surgery, at 3 h after resection of liver, at 24 h after resection of liver and at post operative day 2, and subsequntly analyzed for the above mentioned substances. Routine labs will be monitored until patient is discharged from hospital. During surgery, hemodynamic parameters will be monitored by Picco calculations. Urine output and blood loss will be registred.

ELIGIBILITY:
Inclusion Criteria:

ASA I-III Patient has given informed consent to participate in study.

Exclusion Criteria:

preoperative kidney failure (E-GFR >30), current infection treatment with corticosteroids coagulopathy surgical or anatomical conditions that makes patient unsuitable for participation (for example reoperation, need of vascular bypass, single tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for open liver resection, ASA class I-III.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Ischemic Intestinal Damage | from day of surgery until 24-48 hours postoperatively
  rise in IFABP in nanograms/ml,
Kidney injury | from day of surgery and approximately 1 week onwards
  as described by KDIGO (Kidney Disease Improving Global Outcomes) criteria
Intestinal Bacterial Transloction | from day of surgery until 24-48 hours postoperatively
  Rise in D-lactate in micromol/ml
Kidney injury | from day of surgery until 24-48 hours postoperatively
  proenkephaline increase in pico mol/l
Kidney injury | from day of surgery until 24-48 hours postoperatively
  NAG units/g increase in urine.

SECONDARY OUTCOMES:
Description of Inflammatory Response | from day of surgery and approximately 1 week onwards
  Changes in MCP-1, SDF-1, IL-1beta, TNF-alfa, IL-6, IL-8, IL-10 and HMBG-1, in blood samples obtained during and after heptaic surgery

OTHER OUTCOMES:
blood loss | from day of surgery and approximately 1 week onwards
  need of transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, MD, PhD, professor, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- SahlgrenskaUH, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No